CLINICAL TRIAL: NCT00373737
Title: Microarray Analysis of Gene Expression in Liver Tumors
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Samuel So, Stanford University School of Medicine
Other Study IDs: HEP0005; 76710; HEP0005; NCT00373737
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — liver tumor

SUMMARY:
This study aims to study the gene expression profiles of liver tumors to help us understand their biology, and to find new tumor and treatment markers for liver cancer.

DETAILED DESCRIPTION:
The purpose of this research is to study of the biologic features of liver tissue (by studying their gene expression profiles), so that we can increase our understanding of the processes involved in liver cancer development and growth. This may allow us to identify more effective ways of diagnosing, treating, and predicting the outcome of patients with liver cancer.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria:

* Patients with liver tumors undergoing partial liver resection, open liver biopsy, and patients undergoing liver transplantation with or without liver tumors at Stanford University
* Patients older than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver tumors undergoing partial liver resection, open liver biopsy, and patients undergoing liver transplantation with or without liver tumors at Stanford University
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 1999-05; Primary Completion 2008-04 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel So, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States